CLINICAL TRIAL: NCT03602131
Title: Chidamide Combined With Cladribine/Gemcitabine/Busulfan (ChiCGB) With Autologous Stem-Cell Transplantation in High-risk Hodgkin and Non-Hodgkin Lymphoma
Brief Title: Chidamide Combined With Clad/Gem/Bu With AutoSCT in High Risk Hodgkin & Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCGB-HR lymphomas
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: Chidamide; autologous stem cell transplantation
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cladribine; Gemcitabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ChiCGB (Experimental): Treated with chidamide, cladribine, gemcitabine and busulfan(ChiCGB) therapy followed by autologous hematopoietic stem cell transplantation.
  Interventions: Drug: Chidamide; Drug: Cladribine; Drug: gemcitabine; Drug: Busulfan; Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Chidamide — 30 mg oral twice weekly for 2 weeks
Drug: Cladribine — 6 mg/m2 intravenously once daily for 5 days
Drug: gemcitabine — 2500 mg/m2 intravenously twice weekly for 1 week
Drug: Busulfan — 3.2 mg/kg intravenously once daily for 4 days
Procedure: Autologous hematopoietic stem cell transplantation — autologous hematopoietic stem cells infusion after ChiCGB chemotherapy

SUMMARY:
This study is to explore the efficacy and safety of ChiCGB conditioning therapy in patients with high-risk Hodgkin and non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary refractory or recurrent diffuse large B cell lymphoma, mantle cell lymphoma, peripheral T cell lymphomas, Hodgkin lymphomas that do not qualify for treatment protocols of higher priority.
* Relapsed patients should respond to 2nd or 3rd line salvage chemotherapy and attain at least partial response before recruitment.
* Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min and/or serum creatinine </= 1.8 mg/dL.
* Adequate hepatic function, as defined by serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) </= 3 x upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 x upper limit of normal.
* Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) >/= 50% of expected corrected for hemoglobin.
* Adequate cardiac function with left ventricular ejection fraction >/= 50%. No uncontrolled arrhythmias or symptomatic cardiac disease.
* Performance status 0-1. 10. Negative Beta diffusing capacity of the lung for carbon monoxide (HCG) text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

* Central nervous system lymphoma
* Patients relapsed after autologous stem cell transplantation
* Bone marrow was involved by lymphoma
* Patients with active hepatitis B or C(HBV DNA >/=10,000 copies/mL).
* Active infection requiring parenteral antibiotics
* HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and a normal cluster of differentiation 4 (CD4) counts
* Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
* Patients with a corrected QT interval(QTc) longer than 500 ms

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival | 2 years from recruitment

SECONDARY OUTCOMES:
2-year overall survival | 2 years from recruitment
Treatment related mortality | 2 years from recruitment
non-hematologic adverse events | 2 years from recruitment